CLINICAL TRIAL: NCT06081114
Title: Micronutrient Dose Response (MiNDR) Study in Bangladesh
Brief Title: Micronutrient Dose Response Study in Bangladesh
Acronym: MiNDR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: International Center for Diarrheal Disease Research, Bangladesh (icddr,b) (Unknown); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: INV-033628; IRB00022171 (Other: JHSPH IRB)
Record Dates: First submitted 2023-09-21; First posted 2023-10-13 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Micronutrient Status
Keywords: Pregnancy; Micronutrients; Energy; Supplements; Biochemical indicators; protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MNs - Placebo (Placebo Comparator): Placebo powder, daily in the form of a powdered flavored drink. Plus, a daily fortified balanced energy and protein food supplement containing 400 kcals and 14 g of protein and 1 recommended daily allowance (RDA) of 18 micronutrients will be given daily including 90 ug of vitamin K, 400 ug of folic acid, 1 mg of copper and 500 mg of calcium
  Interventions: Dietary Supplement: Micronutrient Supplement
- MNs - Level 1 (Active Comparator): Dose 1 of micronutrients (MNs) listed provided daily in the form of a powdered drink.
  Micronutrients:
  Vitamin A -0.355 mg Vitamin D - 0.02 mg Vitamin E - 34 mg Vitamin B1 - 1.4 mg Vitamin B2 - 1.4 mg Vitamin B3 - 17 mg Vitamin B6 - 2.1 mg Vitamin B12 - 0.0034 mg Vitamin C - 20 mg Selenium - 0.035 mg Choline - 550 mg Pantothenic acid - 7mg Biotin - 0.035 mg Potassium - 1000 mg Manganese - 2.6 mg Magnesium - 145 mg Plus, a daily fortified balanced energy and protein supplement containing 400 kcals and 14 g of protein and 1 RDA of 18 micronutrients will be given simultaneously including 90 ug of vitamin K, 400 ug of folic acid, 1 mg of Copper and 500 mg of calcium
  Interventions: Dietary Supplement: Micronutrient Supplement
- MNs - Level 2 (Active Comparator): Dose 2 of micronutrients listed below provided daily in the form of a powdered flavored drink.
  Micronutrients:
  Vitamin A -0.93 mg Vitamin D - 0.04 mg Vitamin E - 109 mg Vitamin B1 - 2.8 mg Vitamin B2 - 2.8 mg Vitamin B3 - 47 mg Vitamin B6 - 4.1 mg Vitamin B12 - 0.0094 mg Vitamin C - 20 mg Iron - 10 mg Zinc - 5 mg Selenium - 0.135 mg Choline - 750 mg Pantothenic acid - 7mg Biotin - 0.035 mg Potassium - 1000 mg Manganese - 2.6 mg Magnesium - 145 mg Plus, a daily fortified balanced energy and protein food supplement containing 400 kcals and 14 g of protein and 1 RDA of 18 micronutrients will be given daily including 90 ug of vitamin K, 400 ug of folic acid, 1 mg of copper and 500 mg of calcium
  Interventions: Dietary Supplement: Micronutrient Supplement
- MNs - Level 3 (Active Comparator): Dose 3 of micronutrients listed below provided daily in the form of a powdered drink.
  Micronutrients:
  Vitamin A - 1.48 mg Vitamin D - 0.06 mg Vitamin E - 184 mg Vitamin B1 - 4.2 mg Vitamin B2 - 4.2 mg Vitamin B3 - 82 mg Vitamin B6 - 8.1 mg Vitamin B12 - 0.0154 mg Vitamin C - 20 mg Iron - 10 mg Zinc - 5 mg Selenium - 0.235 mg Choline - 900 mg Pantothenic acid - 7mg Biotin - 0.035 mg Potassium - 1000 mg Manganese - 2.6 mg Magnesium - 145 mg Plus, a daily fortified balanced energy and protein food supplement containing 400 kcals and 14 g of protein and 1 RDA of 18 micronutrients will be given daily including 90 ug of vitamin K, 400 ug of folic acid, 1 mg of copper and 500 mg of calcium
  Interventions: Dietary Supplement: Micronutrient Supplement

INTERVENTIONS:
Dietary Supplement: Micronutrient Supplement — A packaged food supplement providing calories and protein and fortified with micronutrients provided at an approximate RDA.
  Other Names: Balanced Energy and Protein Supplement (BEP)

SUMMARY:
The recommended daily amounts of vitamins and minerals, referred to as micronutrients, are based on data from high income settings and for healthy populations do not fully correct nutritional deficiencies in undernourished settings. This study will determine the minimum acceptable doses across a range of nutrients at which sufficiency is achieved with supplementation using biochemical indicators of nutritional status in non-pregnant (non-lactating) women of reproductive age and pregnant women in Bangladesh. In this double-masked randomized controlled trial, a dose response study will be undertaken using increasing levels of doses provided as supplements to women (pregnant or non-pregnant) with nutritional indicators as outcomes.

DETAILED DESCRIPTION:
The primary aims of the study are to:

1. To characterize the time-course of in vivo exposures (dose response) of several micronutrients in pregnant and non-pregnant and non-lactating women of reproductive age (WRA) in a real-life situation.
2. To characterize any clinically meaningful prognostic factors that can explain the between-subject variability.
3. To investigate whether the micronutrients follow dose-proportional pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

Either

* Women (non-pregnant and non-lactating) and not planning a pregnancy in the next 6 months

OR

* Pregnant women (gestational age at enrollment of 12-14 weeks)

Exclusion Criteria:

* Eligible women not consenting to participate
* Based on point-of-care clinical indicators after enrollment and prior to starting the intervention that is indicative of pre-existing liver or kidney conditions and severe anemia

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 643 (Actual)
Dates: Start 2023-10-22 (Actual); Primary Completion 2025-09-22 (Actual); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in vitamin A status | Baseline, midline, end-line, up to 1 month post-partum (Pregnant women). Baseline, midline, end-line, up to 3 months (non-pregnant women)
  Plasma retinol (μmol/L), retinyl esters (μmol/L), and serum retinol binding protein (μmol/L)
  For women in reproductive age, these biomarkers will be measured at baseline, midline (1.5 months), and end-line (3 months). For pregnant women, the biomarkers will be measured at baseline (10-12 weeks of gestation), mid-pregnancy (22 weeks or 30 weeks of gestation), late pregnancy (36 weeks of gestation), and 1 month postpartum.
Change in vitamin D status | Baseline, midline, end-line, up to 1 month post-partum (Pregnant women). Baseline, midline, end-line, up to 3 months (non-pregnant women)
  Serum 25(hydroxy)D (nmol/L)
  For women in reproductive age, these biomarkers will be measured at baseline, midline (1.5 months), and end-line (3 months). For pregnant women, the biomarkers will be measured at baseline (10-12 weeks of gestation), mid-pregnancy (22 weeks or 30 weeks of gestation), late pregnancy (36 weeks of gestation), and 1 month postpartum.
Change in vitamin E status | Baseline, midline, end-line, up to 1 month post-partum (Pregnant women). Baseline, midline, end-line, up to 3 months (non-pregnant women)
  Plasma α and γ tocopherol (μmol/L)
  For women in reproductive age, these biomarkers will be measured at baseline, midline (1.5 months), and end-line (3 months). For pregnant women, the biomarkers will be measured at baseline (10-12 weeks of gestation), mid-pregnancy (22 weeks or 30 weeks of gestation), late pregnancy (36 weeks of gestation), and 1 month postpartum.
Change in B-vitamin static indicators | Baseline, midline, end-line, up to 1 month post-partum (Pregnant women). Baseline, midline, end-line, up to 3 months (non-pregnant women)
  Vitamin B12 (plasma homocysteine, methylmalonic acid, and holo-transcobalamin, and serum B12); Folic acid (serum folate, and whole blood folate); Vitamin B1 (urinary B1 excretion), Vitamin B2 (urinary B2 excretion), Vitamin B3 (urinary N-methylnicotinamide and 2-pyridone), Vitamin B6 (plasma pyridoxal 5' phosphate and other B6 vitamers, urinary B6 excretion).
  All the indicators will be expressed as pg/ml.
  For women in reproductive age, these biomarkers will be measured at baseline, midline (1.5 months), and end-line (3 months). For pregnant women, the biomarkers will be measured at baseline (10-12 weeks of gestation), mid-pregnancy (22 weeks or 30 weeks of gestation), late pregnancy (36 weeks of gestation), and 1 month postpartum.
Change in B-vitamin enzymatic activity | Baseline, midline, end-line, up to 1 month post-partum (Pregnant women). Baseline, midline, end-line, up to 3 months (non-pregnant women)
  Vitamin B1 (erythrocyte transketolase activity), Vitamin B2 (erythrocyte Glutathione reductase activity, urinary B2 excretion), Vitamin B3 (erythrocyte nicotinamide adenine dinucleotide (NAD) and NAD/nicotinamide-adenine dinucleotide phosphate (NADP) ratio.
  All the indicators will be presented as ratio or activity coefficient.
  For women in reproductive age, these biomarkers will be measured at baseline, midline (1.5 months), and end-line (3 months). For pregnant women, the biomarkers will be measured at baseline (10-12 weeks of gestation), mid-pregnancy (22 weeks or 30 weeks of gestation), late pregnancy (36 weeks of gestation), and 1 month postpartum.
Change in iron status | Baseline, midline, end-line, up to 1 month post-partum (Pregnant women). Baseline, midline, end-line, up to 3 months (non-pregnant women)
  Serum ferritin and soluble transferrin receptor (μg/L)
  For women in reproductive age, these biomarkers will be measured at baseline, midline (1.5 months), and end-line (3 months). For pregnant women, the biomarkers will be measured at baseline (10-12 weeks of gestation), mid-pregnancy (22 weeks or 30 weeks of gestation), late pregnancy (36 weeks of gestation), and 1 month postpartum.
Change in iodine status | Baseline, midline, end-line, up to 1 month post-partum (Pregnant women). Baseline, midline, end-line, up to 3 months (non-pregnant women)
  Urinary iodine (μg/L), and thyroglobulin (μg/L)
  For women in reproductive age, these biomarkers will be measured at baseline, midline (1.5 months), and end-line (3 months). For pregnant women, the biomarkers will be measured at baseline (10-12 weeks of gestation), mid-pregnancy (22 weeks or 30 weeks of gestation), late pregnancy (36 weeks of gestation), and 1 month postpartum.
Change in selenium static indicator | Baseline, midline, end-line, up to 1 month post-partum (Pregnant women). Baseline, midline, end-line, up to 3 months (non-pregnant women)
  Serum selenium (μg/L)
  For women in reproductive age, these biomarkers will be measured at baseline, midline (1.5 months), and end-line (3 months). For pregnant women, the biomarkers will be measured at baseline (10-12 weeks of gestation), mid-pregnancy (22 weeks or 30 weeks of gestation), late pregnancy (36 weeks of gestation), and 1 month postpartum.
Change in selenium enzymatic indicator | Baseline, midline, end-line, up to 1 month post-partum (Pregnant women). Baseline, midline, end-line, up to 3 months (non-pregnant women)
  Plasma Glutathione peroxidase-3 (U/L)
  For women in reproductive age, these biomarkers will be measured at baseline, midline (1.5 months), and end-line (3 months). For pregnant women, the biomarkers will be measured at baseline (10-12 weeks of gestation), mid-pregnancy (22 weeks or 30 weeks of gestation), late pregnancy (36 weeks of gestation), and 1 month postpartum.
Change in zinc status | Baseline, midline, end-line, up to 1 month post-partum (Pregnant women). Baseline, midline, end-line, up to 3 months (non-pregnant women)
  Serum Zinc (μg/L)
  For women in reproductive age, these biomarkers will be measured at baseline, midline (1.5 months), and end-line (3 months). For pregnant women, the biomarkers will be measured at baseline (10-12 weeks of gestation), mid-pregnancy (22 weeks or 30 weeks of gestation), late pregnancy (36 weeks of gestation), and 1 month postpartum.

SECONDARY OUTCOMES:
Changes in inflammation | Baseline, midline, end-line, up to 1 month post-partum (Pregnant women). Baseline, midline, end-line, up to 3 months (non-pregnant women)
  Serum Alpha glycoprotein (AGP) and plasma C-reactive protein (CRP). These will be expressed as mg/L.
  For women in reproductive age, these biomarkers will be measured at baseline, midline (1.5 months), and end-line (3 months). For pregnant women, the biomarkers will be measured at baseline (10-12 weeks of gestation), mid-pregnancy (22 weeks or 30 weeks of gestation), late pregnancy (36 weeks of gestation), and 1 month postpartum.
Change in hormonal markers | Baseline, midline, end-line, up to 1 month post-partum (Pregnant women). Baseline, midline, end-line, up to 3 months (non-pregnant women)
  Plasma hepcidin (μg/L), erythropoietin (μg/L), and serum parathyroid hormone (μg/L)
  For women in reproductive age, these biomarkers will be measured at baseline, midline (1.5 months), and end-line (3 months). For pregnant women, the biomarkers will be measured at baseline (10-12 weeks of gestation), mid-pregnancy (22 weeks or 30 weeks of gestation), late pregnancy (36 weeks of gestation), and 1 month postpartum.
Change in clinical markers of liver enzymes | Baseline, midline, end-line, up to 1 month post-partum (Pregnant women). Baseline, midline, end-line, up to 3 months (non-pregnant women)
  Plasma alanine transaminase (U/L), and Aspartate aminotransferase (U/L)
  For women in reproductive age, these biomarkers will be measured at baseline, midline (1.5 months), and end-line (3 months). For pregnant women, the biomarkers will be measured at baseline (10-12 weeks of gestation), mid-pregnancy (22 weeks or 30 weeks of gestation), late pregnancy (36 weeks of gestation), and 1 month postpartum.
Change in clinical markers of lipid profile | Baseline, midline, end-line, up to 1 month post-partum (Pregnant women). Baseline, midline, end-line, up to 3 months (non-pregnant women)
  Plasma triglyceride, total cholesterol, high density lipoprotein, low density lipoprotein. These will be expressed as mg/dL.
  For women in reproductive age, these biomarkers will be measured at baseline, midline (1.5 months), and end-line (3 months). For pregnant women, the biomarkers will be measured at baseline (10-12 weeks of gestation), mid-pregnancy (22 weeks or 30 weeks of gestation), late pregnancy (36 weeks of gestation), and 1 month postpartum.
Change in clinical markers of renal function | Baseline, midline, end-line, up to 1 month post-partum (Pregnant women). Baseline, midline, end-line, up to 3 months (non-pregnant women)
  Plasma creatinine (mg/dL), and blood urea nitrogen (mg/dL)
  For women in reproductive age, these biomarkers will be measured at baseline, midline (1.5 months), and end-line (3 months). For pregnant women, the biomarkers will be measured at baseline (10-12 weeks of gestation), mid-pregnancy (22 weeks or 30 weeks of gestation), late pregnancy (36 weeks of gestation), and 1 month postpartum.
Change in clinical markers of electrolytes | Baseline, midline, end-line, up to 1 month post-partum (Pregnant women). Baseline, midline, end-line, up to 3 months (non-pregnant women)
  Plasma sodium, calcium, potassium, and chloride. These will be expressed as mmol/L.
  For women in reproductive age, these biomarkers will be measured at baseline, midline (1.5 months), and end-line (3 months). For pregnant women, the biomarkers will be measured at baseline (10-12 weeks of gestation), mid-pregnancy (22 weeks or 30 weeks of gestation), late pregnancy (36 weeks of gestation), and 1 month postpartum.
Change in glucose | Baseline, midline, end-line, up to 1 month post-partum (Pregnant women). Baseline, midline, end-line, up to 3 months (non-pregnant women)
  Plasma glucose (mg/dL)
  For women in reproductive age, these biomarkers will be measured at baseline, midline (1.5 months), and end-line (3 months). For pregnant women, the biomarkers will be measured at baseline (10-12 weeks of gestation), mid-pregnancy (22 weeks or 30 weeks of gestation), late pregnancy (36 weeks of gestation), and 1 month postpartum.
Change in hemoglobin | Baseline, midline, end-line, up to 1 month post-partum (Pregnant women). Baseline, midline, end-line, up to 3 months (non-pregnant women)
  Whole blood hemoglobin (g/L)
  For women in reproductive age, these biomarkers will be measured at baseline, midline (1.5 months), and end-line (3 months). For pregnant women, the biomarkers will be measured at baseline (10-12 weeks of gestation), mid-pregnancy (22 weeks or 30 weeks of gestation), late pregnancy (36 weeks of gestation), and 1 month postpartum.
Change in serum minerals | Baseline, midline, end-line, up to 1 month post-partum (Pregnant women). Baseline, midline, end-line, up to 3 months (non-pregnant women)
  Serum copper, manganese, magnesium, phosphorus, and iron. These will be expressed as μg/L.
  For women in reproductive age, these biomarkers will be measured at baseline, midline (1.5 months), and end-line (3 months). For pregnant women, the biomarkers will be measured at baseline (10-12 weeks of gestation), mid-pregnancy (22 weeks or 30 weeks of gestation), late pregnancy (36 weeks of gestation), and 1 month postpartum.
Change in bone turnover biomarker | Baseline, midline, end-line, up to 1 month post-partum (Pregnant women). Baseline, midline, end-line, up to 3 months (non-pregnant women)
  Pyrilinks-D urine test (nmol/L)
  For women in reproductive age, these biomarkers will be measured at baseline, midline (1.5 months), and end-line (3 months). For pregnant women, the biomarkers will be measured at baseline (10-12 weeks of gestation), mid-pregnancy (22 weeks or 30 weeks of gestation), late pregnancy (36 weeks of gestation), and 1 month postpartum.
Change in urinary metabolite of vitamin E | Baseline, midline, end-line, up to 1 month post-partum (Pregnant women). Baseline, midline, end-line, up to 3 months (non-pregnant women)
  Urinary alpha-carboxy ethyl hydroxy chromanol (nmol/L) will be measured only in pregnancy.
  For pregnant women, the biomarkers will be measured at baseline (10-12 weeks of gestation), mid-pregnancy (22 weeks or 30 weeks of gestation), late pregnancy (36 weeks of gestation), and 1 month postpartum.

OTHER OUTCOMES:
Number of participants with side effects | Weekly from enrollment up to 1 month postpartum for pregnant women. Weekly from enrollment up to 3 months for non-pregnant women
  We will report the number of participants who experience any of the following side effects; Nausea, vomiting, fatigue, headache, hemorrhage, blurred vision, rash, tingling sensation in the extremities, brittleness of nail/hair, dark stool or fishy body odor.
Breastmilk Vitamin A concentration | 1 month postpartum
  Retinol and retinyl esters will be measured by ultra-performance liquid chromatography (UPLC). These will be expressed as μg/L.
Breastmilk Vitamin E concentration | 1 month postpartum
  Plasma α and γ tocopherol will be measured by ultra-performance liquid chromatography (UPLC). These will be expressed as μg/L.
Breastmilk B vitamin concentration | 1 month postpartum
  Vitamin B12, Vitamin B1, B2 and B6 vitamers will be measured by ultra-performance liquid chromatography (UPLC). These will be expressed as μg/L.
Breastmilk mineral concentration | 1 month postpartum
  Zinc, selenium, copper, manganese, magnesium, phosphorus will be measured by Inductively coupled plasma mass spectrometry (ICP-MS). These will be expressed as μg/L.
Change in gut microbiome composition | Baseline, end-line up to 36 wks of gestation in pregnancy (Pregnant women). Baseline, end-line up to 3 months (non-pregnant women)
  Measured by changes in bacterial 16S ribosomal ribonucleic acid gene sequencing (16S RNA) and multigenomic sequencing
  For women in reproductive age, gut microbiome composition will be measured at baseline, and end-line (3 months). For pregnant women, gut microbiome composition will be measured at baseline (10-12 weeks of gestation), and late pregnancy (36 weeks of gestation).
Frequency of neonatal deaths across study arms | Birth to 28 days of life
  Number of deaths between 0-28 days
Frequency of stillbirths across study arms | At birth
  Number of stillbirths
Frequency of low birth weight infants across study arms | At birth
  Low birth weight will be defined as birth weight (within <72 h) less than 2500 g
Frequency of preterm birth across study arms | At birth
  Preterm birth will be defined as babies born alive before 37 weeks of pregnancy are completed
Frequency of gross congenital defects across study arms | At birth
  Any congenital gross malformations at birth that can be identified by physical examination
Frequency of neonatal morbidity across study arms | At 1 month of age
  Will report number of infants experiencing any of the following; fever, cough, cold, difficulty in breathing or diarrhoea.
Change in infant gut microbiome composition, functional profile and maturation | 3-6 months and 6-9 months of infant age
  Measured by metagenomic sequencing of total fecal DNA
Change in human milk oligosaccharide composition | 1 month, 3-6 months and 6-9 months of infant age
  Measured by quantification of the 19 most abundant HMOs - representing 95% of total HMO concentration in milk and all structural features using HPLC with flouresence detection. We aim to examine the impact of the micronutrient interventions on HMOs in human milk.
Infant length-for-age z-score | 3-6 months and 6-9 months of infant age
  Anthropometry taken using length board. We aim to examine difference in infant length-for-age z-score by intervention arm as well effect modification by microbiota maturity on stunting.
Infant weight-for-length z-score | 3-6 months and 6-9 months of infant age
  Measured using a pediatric digital scale. We will examine the difference in WLZ score by intervention arm and effect modification of microbiota maturity on wasting (WLZ< -2)

CONTACTS AND LOCATIONS:
Overall Officials: Parul Chrisian, DrPH, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- JiVitA Project, Rangpur City, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Siddiqua TJ, Schulze KJ, Hasan ST, Ahsan KB, Bandyopadhyay S, Zavala E, Ali H, Haque R, Sujan HM, Rahman MH, Baker S, Stephenson KK, Ge X, Gough EK, Langevin B, Wu LSF, Dyer B, Roy AK, Jubair M, Nishan AA, Rosenblum M, Gopalakrishnan M, Kraemer K, Erchick DJ, Ahmed T, Christian P. Micronutrient dose response (MiNDR) study among women of reproductive age and pregnant women in rural Bangladesh: study protocol for double-blind, randomised, controlled trials. BMJ Open. 2025 Jan 4;15(1):e090108. doi: 10.1136/bmjopen-2024-090108. PMID 39755576
- See also: Trial protocol — https://pubmed.ncbi.nlm.nih.gov/39755576/